CLINICAL TRIAL: NCT03440671
Title: A Multicenter, Double-Blind, Randomized, Parallel, Active-controlled, Non-inferiority, Phase 3 Clinical Trial to Compare the Efficacy and Safety Study of Hutox Versus Botox® in Subject With Moderate to Severe Glabellar Lines
Brief Title: The Safety and Efficacy Study of Hutox Versus Botox® in Subject With Moderate to Severe Glabellar Lines
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HU-014_P3
Record Dates: First submitted 2018-01-11; First posted 2018-02-22 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Glabellar Frown Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hutox Inj (Experimental): Hutox Inj was given an injection to 5 glabellar lines each 4 U/0.1ml (Total 20 U/0.5ml, IM)
  Interventions: Biological: Hutox Inj
- Botox Inj (Active Comparator): Botox Inj was given an injection to 5 glabellar lines each 4 U/0.1ml (Total 20 U/0.5ml, IM)
  Interventions: Biological: Botox Inj

INTERVENTIONS:
Biological: Hutox Inj — Hutox Inj(Clostridium botulinum type A)
  Arms: Hutox Inj
Biological: Botox Inj — Botox Inj(Clostridium botulinum type A)
  Arms: Botox Inj

SUMMARY:
A Phase Ⅲ Clinical Trial to Compare the Safety and Efficacy of Hutox versus Botox® in Subject with Moderate to Severe Glabellar Lines

ELIGIBILITY:
Inclusion Criteria:

* Facial Wrinkle Scale (FWS) score > 2 when Subject knits brow extremely

Exclusion Criteria:

* Volunteer who has history of any diseases following. (myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis etc.)
* From screening, Subject who get a plastic Surgery including fascioplasty, Prosthesis implantation within 6 Weeks
* Subject who takes a medication including skeletal muscle relaxants, Aminoglycoside, lincomycin, anticholinergic drug, benzodiazepine, benzamide etc
* Subject who takes a medication including anticoagulant, antithrombotic drug except low dose aspirin (below 325 mg/day)
* Any condition that, in the view of the investigator, would interfere with study participation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
FWS(Facial Wrinkle Severity) Improvement at glabellar line | 4 Weeks
  Change from Baseline of Glabellar Lines improvement rate(Frown)

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Seongnam-si, Gyeonggi-do, South Korea